CLINICAL TRIAL: NCT03475264
Title: MRI of Lung Structure and Function in Preterm Children
Status: Terminated | Type: Observational
Why Stopped: Recruitment and Funding challenges
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Giles Santyr, Senior Scientist, The Hospital for Sick Children
Other Study IDs: 1000055897
Record Dates: First submitted 2018-02-06; First posted 2018-03-23 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Lung MRI, Bronchopulmonary Dysplasia, hyperpolarized xenon,
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy: Healthy Participants
  Interventions: Diagnostic Test: Lung MRI
- BPD cohort: Participants born prematurely with a diagnosis of BPD
  Interventions: Diagnostic Test: Lung MRI
- Non-BPD cohort: Participants born prematurely without a diagnosis of BPD
  Interventions: Diagnostic Test: Lung MRI

INTERVENTIONS:
Diagnostic Test: Lung MRI — Participants will be undergoing hyperpolarized xenon and proton lung MRI

SUMMARY:
The MRI tools developed by the investigators are well positioned for assessing regional changes in lung structure and function in preterm children with bronchopulmonary dysplasia (BPD), in which airway limitation similar to asthma, alveolar simplification similar to emphysema and pulmonary vascular stunting are expected. To the investigator's knowledge, the combination of ultra short echo time (UTE) proton, pulmonary vascular proton and hyperpolarized 129Xe MRI have not yet been explored in BPD, either clinically or preclinically. The investigators propose that a comprehensive MRI examination may be useful from a diagnostic perspective, MRI of preterm children without BPD may reveal changes which are otherwise clinically 'silent' yet still place children at risk for future chronic lung disease in later life.

DETAILED DESCRIPTION:
Briefly, at the beginning of an approximate three hour study visit, the qualified investigator (QI) / delegate will explain the study procedure to the participants and the participants will have an opportunity to ask questions regarding the study procedure. Following the explanation of the study, written informed consent will be collected at the beginning of visit 1. Participants who are deemed unable to provide consent will be provided an assent form and consent will be acquired from their parents/ legal guardians. During the study visit, participants will undergo: 1) brief medical history and clinical examination including questionnaires, 2) full pulmonary function tests, lung clearance testing (LCI), forced oscillation technique (FoT) and exercise testing, 3) proton MRI, 4) spin-density and/or diffusion-weighted 129Xe MRI, 5) Multiple-breath washout imaging. Qualified research team members will perform a clinical examination on the participant to record their vital statistics like age, gender, height, weight, heart rate, respiratory rate, oral temperature and blood pressure. The QI/delegate, during a brief conversation with the participant, will collect relevant medical history from the participant to make sure the participant meets all the inclusion/exclusion criteria for the study. The QI will also make sure that the participant understands the study procedure and is willing to participate in the study. Based on the clinical examination results, medical history and the pulmonary function test results, the QI/delegate will determine if all the inclusion/exclusion criteria are met to proceed with the MRI part of the study visit.

ELIGIBILITY:
Inclusion Criteria:

- Children born pre-term at less than 28 weeks' gestation, currently aged 6-9 years, with and without BPD will be included.

For the preterm non-BPD cohort, inclusion will include

* no requirement of supplementary oxygen beyond 28 days from birth. For the BPD preterm cohort, inclusion criteria will include
* need for oxygen at 36 weeks' postmenstrual age, which includes those with moderate-severe disease .

For the healthy cohort, inclusion will include

-absence of any diagnosed pulmonary disease and term birth.

Exclusion Criteria: Children with

* known interstitial lung disease, congenital lung anomalies, cystic fibrosis, ciliary dysfunction, immunodeficiency, neuromuscular disease or structural heart disease, which may have associated pulmonary function tests (PFT) and/or MRI findings;
* genetic syndromes which may have other associated structural lung anomalies;
* any contraindications for MRI
* severe neurosensory deficits which would prevent test completion;
* viral or bacterial respiratory infection within 6 weeks will be excluded. For all three groups (healthy, preterm non-BPD and preterm BPD), we will exclude
* those with congenital lung disease (i.e. Congenital diaphragmatic hernia (CDH), lung cysts) or non BPD acquired chronic lung disease as defined by need for any routine supplementary oxygen
* if the participant has an MRI incompatible device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bio prosthetic, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants).

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy volunteers will be selected from the general population and the BPD and non-BPD cohorts will be selected from patients from clinics seen at the Hospital for Sick Children, Toronto
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
MRI ventilation and 1H MRI thoracic cavity volume and tissue density | 2 years
  Ventilation defect percent (VDP) (%) will be generated for whole lung and individual lung slices using manual or semi-automated segmentation. For proton (1H) thoracic cavity images, the thoracic cavity volume (TCV) will be calculated by manual or semi-automated segmentation.

SECONDARY OUTCOMES:
Apparent Diffusion Coefficients (ADC) and ADC maps | 2 years
  Diffusion weighted images from each visit will be reviewed and compared with the proton anatomical images. Mean, whole lung, and center slice ADC (and standard deviation) will be calculated and recorded.
Multiple breath washout testing: | 2 years
  VDP will be calculated as described above based on the first image data set prior to wash-out breaths. A pixel-by-pixel fit of images as a function of washout breath number will then be used to calculate the fractional ventilation map defined as the volume of expired gas leaving a volume divided by its end-inspiratory volume.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers outside of the institutions